CLINICAL TRIAL: NCT06883409
Title: Efficiency of Laparoscopic Interval Cytoreductive Surgery After Neoadjuvant Chemotherapy in Patients With Stage III and IV Epithelial Ovarian Cancer
Brief Title: Laparoscopic Interval Cytoreductive Surgery in Advance Ovarian Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Cancerologia de Mexico (Other)
Responsible Party: Principal Investigator, David Isla Ortiz, Head of Department of Gynecological Oncology, None in Three Research Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INCAN MEXICO
Record Dates: First submitted 2025-01-23; First posted 2025-03-19 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Ovarian Neoplasms
Keywords: Minimal invasive surgery; interval debulking surgery; advance ovarian cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Intervention Model Description: A prospective single-arm phase II clinical trial study was conducted. We evaluated the efficacy and complications of interval laparoscopic cytoreduction in patients with COEA after NCT. Patients diagnosed with advanced ovarian carcinoma who received 3 to 4 cycles of NCT using carboplatin/paclitaxel with or without bevacizumab were included. Interval cytoreductive laparoscopic surgery was performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with advance ovarian cancer already treated with NACT and eligible for MIS (Experimental): Were enrolled patients who met the inclusion criteria by receiving 3 to 4 cycles of NACT, with ca 125 up to 200 U/ml, and partial or complete response by image (PET-CT), and subsequently underwent laparoscopic approach.
  Interventions: Procedure: Interval Cytoreduction Surgery

INTERVENTIONS:
Procedure: Interval Cytoreduction Surgery — The procedure started with the cytoreduction of highest complexity (determined at the time of initial inspection), after which, if necessary, the patient underwent a complete hysterectomy, bilateral salpingo-oophorectomy, omentectomy, or partial peritonectomy and excision of any peritoneal implants present. The magnitude of the surgical procedures will be classified as:
  1. Standard surgery: minimal hysterectomy, adnexectomy y omentectomy
  2. Radical Surgery: included resection of the ovaries, of the rectouterine excavation (pouch of Douglas) and or the peritoneum between the bladder and uterus, hysterectomy, rectosigmoid colectomy, and complete omentectomy
  3. Supra-radical Surgery: included other procedures such as splenectomy, diaphragm resection, or other intestinal resection.

SUMMARY:
This is a study that aims to demonstrate the non-inferiority of minimally invasive surgery versus open surgery, as an approach for patients with advanced ovarian cancer who received neoadjuvant chemotherapy, giving them the benefits of laparoscopic surgery. This way they can continue with their complementary treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of epithelial ovarian cancer (all subtypes of epithelial ovarian cancer) in stage III-IV
* Partial and complete response to treatment with QTNA after 3-4 cycles, evaluated by PET-CT imaging study, patients that the functional unit decides to incorporate into the project.
* Ca 125 which will have to be less than 200
* ECOG 0 to 2 without medical contraindication to perform surgery (≤ ASA 2 or ≤ Goldman 2).

Exclusion Criteria:

* Partial response with persistence of ascites or pleural effusion.
* With unresectability criteria (multiple intrahepatic liver metastases, retroperitoneal lymph node conglomerates >2cm above the renal lymph nodes, metastatic disease above the diaphragm, multiple intestinal involvement and mesentery retraction).

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2022-05-19 (Actual); Primary Completion 2024-06-14 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Efficiency of Laparoscopic Interval Cytoreductive Surgery After Neoadjuvant Chemotherapy in Patients with Stage III and IV Epithelial Ovarian Cancer | 1 year
  Efficiency of laparoscopic interval surgery will be evaluated according to percentage of patients who achieved optimal cytoreduction compared to the reported rates in the literature (70 -80%) and the measured frequency of complications during the 30 day postoperative period. Severity of complications will be measured using the Clavien Dindo scale (Grade I: any deviation from the normal post operative course without need for pharmacological treatment - Grade V: death)

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Nacional de Cancerologia, México, Tlalpan, Mexico

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-03-24): https://cdn.clinicaltrials.gov/large-docs/09/NCT06883409/Prot_SAP_001.pdf